CLINICAL TRIAL: NCT00162903
Title: The Role of Nitric Oxide, Endothelin-1, and Inflammatory Mediators in the Patency of Ductus Arteriosus in Preterm Infants
Brief Title: Nitric Oxide, Endothelin-1, and the Patency of Ductus Arteriosus in Preterm Infants
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 26955
Record Dates: First submitted 2005-09-12; First posted 2005-09-13 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2001-10

CONDITIONS: Patent Ductus Arteriosus
Keywords: Preterm infant, Patent ductus arteriosus, Nitric oxide,Endothelin-1
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
BACKGROUND Patent ductus arteriosus (PDA) is a frequent clinical event in preterm infant. The cardiopulmonary functions of these preterm babies may be adversely affected by the patency of ductus arteriosus. Ductal tissues are sensitive to the constricting effect of endothelin-1 and the dilating effect of prostaglandins, inflammatory mediators, and concentration of oxygen.

OBJECTIVE To examine the role of endogenous nitric oxide (NO) and endothelin-1 (ET-1) in the pathogenesis of patent ductus arteriosus of the preterm infants. We hypothesize that the patency of ductus arterious in preterm infants is probably due to inappropriate production of endogenous nitric oxide and the interaction with various inflammatory mediators and prostaglandins, which is different from those of term infants. In addition, the secretion of endothelin is probably decreased. The purpose of this study is to monitor the changes of these substance sequentially, and to evaluate the relationship among endothelin-1, endogenous nitric oxide, and inflammatory mediators in the pathophysiology of patent ductus arteriosus in preterm infants.

METHODS AND MATERIALS

1. Inclusion criteria:

   1. Preterm infants with gestational age less than 32 weeks or birth weight less than 2000 gm.
   2. Informed consent
2. Numbers of study population:

   With 80-100 evaluable infants (40-50 patients in PDA and non-PDA groups, respectively)
3. Blood sample, collecting on day 1,3,7 after regular echocardiographic evaluation, is assessed for inflammatory mediator (IL-8, IL-10), nitric oxide metabolites (nitrite and nitrate), endothelin-1, and cGMP
4. Statistical analysis: Student t-test testing the differences of clinical data, Wilcoxon signed rank test for comparing data obtained between the PDA and non-PDA patients, the PDA patients before and after intravenous indomethacin, and those who are responsive or refractory to the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of the patency of ductus arteriosus

Exclusion Criteria:

* Congenital anomalies

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80
Dates: Start 2002-01; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Wu Shiun Hsieh, M.D, Study Director — National Taiwan University Hospital